CLINICAL TRIAL: NCT06564116
Title: A Randomized, Double-blind, Active Comparator Clinical Trial to Evaluate Safety and Immunogenicity of Thiomersal-free Recombinant Hepatitis E Vaccine (Escherichia Coli) in People Ages 16 Years and Above
Brief Title: Safety and Immunogenicity Study of Thiomersal-free Hepatitis E Vaccine in People Ages 16 Years and Above
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xiamen Innovax Biotech Co., Ltd (Industry)
Collaborators: Center for Disease Control and Prevention, Fujian (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRO-HE-011
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Hepatitis E
Keywords: Hepatitis E; Hepatitis E vaccine; Thiomersal
MeSH Terms: conditions — Hepatitis E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Thiomersal-free hepatitis E vaccine
  Interventions: Biological: Thiomersal-free Recombinant Hepatitis E Vaccine (Escherichia Coli)
- Control Group (Active Comparator): Licensed hepatitis E vaccine
  Interventions: Biological: Recombinant Hepatitis E Vaccine (Escherichia Coli)

INTERVENTIONS:
Biological: Thiomersal-free Recombinant Hepatitis E Vaccine (Escherichia Coli) — Participants would receive 3 doses of thiomersal-free hepatitis E vaccine intramuscularly at month 0, 1 and 6.
  Arms: Test Group
Biological: Recombinant Hepatitis E Vaccine (Escherichia Coli) — Participants would receive 3 doses of licensed hepatitis E vaccine intramuscularly at month 0, 1 and 6
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate the safety and non-inferior immunogenicity of thiomersal-free Recombinant Hepatitis E Vaccine (Escherichia Coli) compared with licensed Recombinant Hepatitis E Vaccine (Escherichia Coli) when administered in participants ages 16 years and above.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, active-comparator study to evaluate the safety and immunogenicity of thiomersal-free Recombinant Hepatitis E Vaccine (Escherichia Coli) in participants ages 16 years and above. Sex (male, female) and age (16-40 years old, 41 years old and above) are used as stratified factors. Participants are randomly assigned in a 1:1 ratio to receive three doses of thiomersal-free hepatitis E vaccine or licensed hepatitis E vaccine intramuscularly at Month 0, 1 and 6. The vaccine safety is assessed from the 1st dose vaccination to 6 months after the last dose vaccination. Serum samples are collected for anti-HEV IgG determination at Month 0 and 7.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 16 years and above when administered with the first dose of vaccine;
2. Axillary temperature is 37.2 ℃ or less;
3. Clinically determined as healthy and eligible for vaccination by the investigators after inquiring about the medical history and relevant physical examinations;
4. Willing to participate in this study and sign informed consent form (ICF). Participants aged 16-17 years should sign ICF jointly by themselves and their guardians;
5. Able to comply with the request of study protocol and complete every visit;
6. Females with negative urine pregnancy test results;
7. Negative serological markers for hepatitis E (HEV-Ab).

Exclusion Criteria:

1. Females who are pregnant or breastfeeding, or planning to be pregnant within the next 8 months;
2. Administration of hepatitis E vaccine before the study;
3. Use of any investigational product or non-registered product (drug or vaccine) within 30 days preceding the first dose of the study vaccine or plan to use during the study period;
4. Long-term (for more than 14 days) use of immunosuppressant, immunoregulation therapy or corticosteroid systemic therapy within 6 months before the first dose of the study vaccine, excluding local treatment ( such as ointment, eye drops, inhalants or nasal sprays);
5. Administration of any immunoglobulin or blood products within 3 months preceding the first dose of the study vaccine, or plan to use during the study period;
6. Administration of any inactivated vaccines within 14 days preceding enrollment (other vaccines besides live-attenuated vaccines, including recombinant vaccines, subunit vaccines, polysaccharide conjugate vaccines, synthetic peptide vaccines, etc ), or live-attenuated vaccines within 28 days preceding enrollment;
7. Had a fever (axillary temperature is 38.0℃ or higher) within 3 days prior to, or any acute illness requiring systemic antibiotics or antiviral treatment within 5 days prior to vaccination;
8. Plan to participate in any other clinical trial during the study period;
9. Immunodeficiency disorders, subjects with primary diseases of important organs, cancer or precancerous lesions, or any immune disease requiring treatment (such as systemic lupus erythematosus, rheumatoid arthritis, any condition resulting in asplenectomy or splenectomy, and other immune diseases that researchers believe may have an impact on the immune response);
10. Have a history of severe allergies, including history of serious adverse events occurring after vaccination, i.e., allergy,urticaria, dyspnea, angioneurotic edema or abdominal pain.
11. Asthma that needed emergency treatment, hospitalization, oral or intravenous corticosteroid to keep stable in the past two years;
12. Complicated with another severe internal disease(such as hypertension, cardiopathy, diabetes and hyperthyroidism etc);
13. Abnromal coagulation function (such as coagulation factor deficiency, coagulation disorders, platelet abnormalities) or coagulopathy diagnosed by the doctor;
14. Epilepsy, excluding febrile seizures under 2 years old, alcoholic seizures within 3 years before abstinence, or simple epilepsy without treatment in the past 3 years;
15. Inability to comply with the study requirement due to psychological conditions, past or present severe mental disorders that have not been well controlled within the past 2 years, accident-causing behavior, or having suicidal tendencies in the past 5 years;
16. Other medical, psychological, social or occupational factors that, according to the investigators' judgment, which are inconsistent with the study protocol or affecting the subjects and/or guardians (trustees) to sign the informed consent;
17. Individuals without civil capacity.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate of anti-HEV IgG at Month 7 | Month 7
  The percentage of participants who had ≥4-fold rise in anti-HEV IgG antibody from baseline to Month 7.
Anti-HEV IgG geometric mean concentration (GMC) at Month 7 | Month 7
  Measure anti-HEV IgG antibody GMC at Month 7.
Adverse events within 0-7 days after each vaccination | Day 7
  Measure percentage of participants reporting adverse events within 0-7 days after each vaccination.
Adverse events within 8-30 days after each vaccination | Day 30
  Measure percentage of participants reporting adverse events within 8-30 days after each vaccination.
Serious adverse events and pregnancy from the 1st dose vaccination to 6 months after the last vaccination | Month 12
  Measure percentage of participants reporting serious adverse events and pregnancy from the 1st dose vaccination to 6 months after the last vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Dongjuan Zhang, Principal Investigator — Center for Disease Control and Prevention, Fujian
Locations (1):
- Youxi County Center for Disease Control and Prevention, Sanming, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li J, Wang X, Zhang D, Xie F, Zhong S, Yu X, Chen S, Huang Q, Wang R, Zhang Q, Zhang D. Safety and immunogenicity of thiomersal-free recombinant hepatitis E vaccine: A randomized, double-blind, active-controlled study. Vaccine. 2025 Aug 30;62:127510. doi: 10.1016/j.vaccine.2025.127510. Epub 2025 Jul 20. PMID 40690851